CLINICAL TRIAL: NCT05860985
Title: Zeiss RESIGHT Disposable Lenses Evaluation Study: Investigator-initiated, Mono-center, Academic, Prospective, Interventional Case Study
Brief Title: Zeiss RESIGHT Disposable Lenses Evaluation Study
Acronym: RESIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: S67415
Record Dates: First submitted 2023-04-13; First posted 2023-05-16 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Retinal Detachment; Macular Pucker; Macular Holes; Vitreomacular Traction
MeSH Terms: conditions — Retinal Detachment; Epiretinal Membrane; Retinal Perforations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Active Comparator): primary vitrectomy surgery for retinal detachment
  Interventions: Device: ZEISS disposable
- group 2 (Active Comparator): macular surgery: pucker, vitreomacular traction or macular hole
  Interventions: Device: ZEISS disposable

INTERVENTIONS:
Device: ZEISS disposable — a comparison will be done between the present lenses used (reusable RESIGHT lenses and disposable Vitreq contact lens) and the new disposable RESIGHT lenses.

SUMMARY:
To evaluate the intra-operative efficacy of a new intra-operative viewing device.

DETAILED DESCRIPTION:
This study is designed to obtain more information on the efficacy of the disposable RESIGHT lenses in routine vitrectomy surgery. This information can lead to adjustments to these surgical lenses to further fine tune a device which can be used by other surgeons.

Theoretically, both the improved lens design and better resistance to fogging should improve the visualization of the retina hence facilitate the surgery, increasing the surgical safety.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
* Patients that are scheduled for primary vitrectomy surgery to treat retinal detachment or macular disease (pucker, macular hole, vitreomacular traction).
* Both vitrectomy-only and combined phaco-vitrectomy surgeries
* General or local anesthesia, or combination

Exclusion Criteria:

* Patient who do not have sufficient command of the Dutch language to read and understand the informed consent form
* Any disorder, which in the investigator's opinion might jeopardise participant's safety or compliance with the CIP.
* Repeat vitrectomy surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Ultra Wide Field lens View Angle evaluation | during surgery
  Ultra Wide Field lens View Angle: scale from 1 (far more indentation) to 5 (far less indentation)
Ultra Wide Field lens Condensation evaluation | during surgery
  Ultra Wide Field lens Condensation: scale from 1 (far more condensation) to 5 (far less condensation)
Wide Angle lens Condensation evaluation | during surgery
  Wide Angle lens Condensation: scale from 1 (far more condensation ) to 5 (far less condensation)
Illumination appearance evaluation | during surgery
  Illumination intensity required during the surgery : scale from 1 (significantly higher) to 5 (significantly lower)
Color appearance evaluation | during surgery
  color appearance during the surgery : scale from 1 (far less natural colors) to 5 (far better natural colors )

CONTACTS AND LOCATIONS:
Overall Officials: Peter Stalmans, PhD, MD, Principal Investigator — UZ Leuven
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Vlaams-Brabant, Belgium

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-07): https://cdn.clinicaltrials.gov/large-docs/85/NCT05860985/Prot_SAP_000.pdf